CLINICAL TRIAL: NCT02669147
Title: A Study to Determine Enzalutamide Long-term Safety and Efficacy After Anti-androgen Therapy for CRPC
Acronym: DELC
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Sponsor
Other Study IDs: TRIGU1517; UMIN000019855 (Other: UMIN-CTR)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Castration Resistant Prostate Cancer (CRPC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective observational study to evaluate effectiveness and safety of Enzalutamide for Castration Resistant Prostate Cancer (CRPC) patients who decided to administer Enzalutamide after anti-androgen therapy.

CRPC Patients who are observed PSA or disease progression after anti-androgen therapy and decided to administrate Enzalutamide will dose the Enzalutamide 160 mg orally once daily and observed the practical treatment. Total research term is for 4 years, consists of 2-year case registration terms and 2-year observational terms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed prostate cancer.
2. Patients who are receiving or received continuous androgen deprivation therapy using both gonadotropin-releasing hormone (GnRH) agonist and antagonist (medical castration), or both testicles removal by surgery (surgical castration).
3. Castration resistant prostate cancer (CRPC) patients who are observed disease progression after castration treatment and implied the treatment resistant.
4. CRPC patients who conducted anti-androgen alternating therapy as shown below 1) and are observed one or more of disease progression shown as below 2) during or after the therapy and decided to administer enzalutamide.

   Note 1) anti-androgen alternating therapy is defined as the therapy of flutamide administration after bicalutamide.

   Note 2) Disease progression criteria during or after anti-androgen alternating therapy

   ① PSA progression during or after anti-androgen alternating therapy: PSA increased more than 25% compare to the lowest test results after initial dose of anti-androgen alternating therapy (flutamide) and the increasing is more than 2ng/ml.

   ②Confirmed disease progression of soft tissue lesion defined as RECIST v1.1.

   ③Confirmed disease progression of bone lesion defined as 2 or more of new appearance of bone lesion on bone scintigraphy.
5. Patients with the Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Patients who have signed written informed consent to participate in this study

Exclusion Criteria:

1. Patients who is administering or have administration history of enzalutamide, abiraterone, docetaxel or cabazitaxel
2. Patients with history of seizure or predisposing disease of seizure
3. Patients with severe liver dysfunction
4. Patients with a previous history of hypersensitivity to any component of drugs which will be administered in this study
5. Patients who considered to be inappropriate for the study participation by the investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRPC patients who are observed PSA or disease progression after anti-androgen therapy and decided to administrate Enzalutamide
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 50 months
  OS is defined as time from date of initial dose until date of death from any cause. In the case of any new chemotherapy added or changed to another treatment to prostate cancer, the conducted date will be applied. When patient is no longer traceable, the final confirmed date as alive will be applied to OS.

SECONDARY OUTCOMES:
Prostate Specific Antigen-progression-free survival (PSA-PFS) | 50 months
  Prostate specific antigen (PSA) progression-free survival is defined as time from date of initial dose until the date of first confirmed PSA progression (an increase in PSA of >= 25% and >= 2 ng/ml above the nadir after initial dose) or date of death from any cause, whichever comes first. In the case of any new chemotherapy added or changed to another treatment to prostate cancer, the conducted date will be applied.
Progression-free survival (PFS) | 50 months
  PFS is defined as time from date of initial dose until the date of first confirmed progression or date of death from any cause, whichever comes first. Progression is defined as followed:① A growth of primary lesion or appearance of neopathy by image diagnosis, aggravation of general condition・PS decrease or noticable weight loss which investigator assess as progression. ②Unmeasurable or difficult to measure lesion which newly appeared or investigator assess as obvious aggravation. ③ In the case of any new chemotherapy added or changed to another treatment to prostate cancer
Time to Treatment Failure (TTTF) | 50 months
  TTTF is defined as time from date of initial dose until the date of any new chemotherapy added or changed to another treatment to prostate cancer.
Time-to-PSA-progression (TTPP) | 50 months
  TTPP is defined as time from date of initial dose until the date of first confirmed PSA progression (an increase in PSA of >= 25% and >= 2 ng/ml above the nadir after initial dose). In the case of any new chemotherapy added or changed to another treatment to prostate cancer, the conducted date will be applied.
PSA response rate | 50 months
  PSA response rate is defined as ratio of patients who have an decrease in PSA of >= 50% above baseline since initial dose.
Time to First Symptomatic Skeletal Events (TTFS) | 50 months
  TTFS is defined as time from date of initial dose until the date of first confirmed skeletal-related event. In the case of any new chemotherapy added or changed to another treatment to prostate cancer, the conducted date will be applied. Symptomatic Skeletal Events (SSE) defined as followed: ・Operation of EBRT External Beam Radiation Therapy (EBRT) to mitigate skeletal events ・New appearance of symptomatic pathological fracture ・Appearance of spinal cord compression ・Orthopedic intervention related to tumor
The state of administration | 2 years
  The state of administration is assessed by Relative Dose Intensity (RDI). RDI is calculated by dosage and dosing period. RDI calculation formula =∑ (daily dosage ×dosing days) / (160mg ×total dosing number of days). ∑ means all total dose which adds up in different dosage. Total number of days mean treatment term of this trial.
Safety assessment | 50 months
  Safety assessment by the incidence and severity of adverse events as assessed by Japanese version of the Common Terminology Criteria for Adverse Events (CTCAE) version 4.00

CONTACTS AND LOCATIONS:
Overall Officials: Norio Nonomura, MD, Ph.D., Study Chair — Osaka University Graduate School Of Medicine, Department of Urology